CLINICAL TRIAL: NCT01844453
Title: Impact of Local Endometrial Injury on Implantation Rates in Fresh Embryo Transfer Cycles
Brief Title: Local Endometrial Injury in Fresh Embryo Transfer Cycles
Acronym: LEI
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Dr. Dan Nayot, B.Sc.; M.Sc.; M.D., McGill University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3216
Record Dates: First submitted 2013-04-29; First posted 2013-05-01 (Estimated); Last update posted 2013-05-01 (Estimated); Status verified 2013-04

CONDITIONS: Infertility
Keywords: Subfertility; Recurrent Implantation Failure
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- Luteal Phase Arm (Experimental): Local Endometrial Injury in mid-luteal phase (cycle day 21-26) prior to the treatment cycle.
  Interventions: Procedure: Endometrial Biopsy
- Proliferative Phase Arm (Experimental): Local Endometrial Injury in early proliferative phase of current treatment cycle (cycle day 2-3).
  Interventions: Procedure: Endometrial Biopsy
- Control Arm (No Intervention): No Local Endometrial Injury will be performed. Patients will undergo a routine fresh IVF treatment cycle.

INTERVENTIONS:
Procedure: Endometrial Biopsy — The Local Endometrial Injury will be performed using the standard technique using a Pipelle sampling catheter in the outpatient department. After a speculum examination is performed and the cervix is well visualized, the Pipelle will be inserted gently through the cervical canal into the uterine cavity and advanced slowly until resistance is noted. At this point the internal piston is withdrawn to create negative suction and the Pipelle is gently maneuvered up and down alongside the uterine cavity wall. The Pipelle catheter is then withdrawn gently and any obtained specimen (uterine lining) will be sent for histopathological examination.
  Other Names: Local Endometrial Injury
  Arms: Luteal Phase Arm; Proliferative Phase Arm

SUMMARY:
The application of in-vitro fertilization (IVF) has provided remarkable opportunities for infertile couple to conceive in the last four decades. Historically IVF was performed for patients with bilateral tubal obstruction, but its use is presently widespread. Although the efficacy of assisted reproductive technology continues to improve, endometrial implantation remains the limiting step towards a successful pregnancy. Reduced endometrial receptivity and embryonic defects are the probable primary causes of implantation failure during IVF(1). Patients with repeated implantation failure despite transferring good-quality embryos continue to be a major dilemma for clinicians and are a topic of great research interest. Barash et al. unintentionally discovered and initially reported that an endometrial biopsy prior to IVF in women who have had one or more implantation failures was associated with an increased clinical pregnancy (66.7% vs 30.3%, p<0.01) and live birth rates 48.9% vs 22.5%, p=0.02) compared to a control group(2). The mechanism by which a local endometrial injury (LEI) may increase the pregnancy rate is still not fully clear. Possible etiologies include its role in promoting a beneficial local inflammatory response, inducing endometrial decidualization, or improving endometrial maturation synchrony (3-6).

Following Barash et al's publication, several randomized controlled studies confirmed their findings (7-11). However, there has been extensive heterogeneity among studies, including the number of biopsies, how the biopsy is performed and the selected patient population. On the other hand all the studies have in common that the endometrial biopsy was performed prior to the start of the IVF cycle.

The optimal timing of an endometrial biopsy with respect to an IVF cycle is unknown. There is reason to suspect that an endometrial biopsy during the follicular phase of an IVF stimulation cycle may improve pregnancy outcomes, although this has not been directly examined. We therefore propose a randomized controlled study to evaluate the impact of an endometrial biopsy on the implantation and pregnancy rate in both the luteal phase prior to the IVF cycle as well as the follicular phase of the concurrent IVF cycles.

DETAILED DESCRIPTION:
HYPOTHESIS

1. Local endometrial injury improves implantation and pregnancy rates
2. Specifically, local endometrial injury during the follicular phase of an IVF cycle improves the implantation and pregnancy rates in comparison to that in the luteal phase prior to ovarian stimulation .

OBJECTIVES Primary objective

•To determine the impact of local endometrial injury on implantation rates in patients undergoing fresh IVF cycles.

Secondary objectives

* To determine the impact of local endometrial injury on pregnancy outcomes (biochemical pregnancy rate, clinical pregnancy rate, miscarriage rate and live birth rate) in patients undergoing fresh IVF cycles.
* To determine the optimal timing for local endometrial injury (mid-luteal phase prior to ovarian stimulation or early follicular phase during ovarian stimulation) to improve pregnancy outcomes.
* To determine if there is a correlation between endometrial biopsy pathology and IVF pregnancy outcomes among patients randomized to local endometrial injury.

STUDY DESIGN The study will be a randomized controlled study (RCT) and consists of patients undergoing fertility treatment with their second fresh IVF cycle, which includes ovarian stimulation with gonadotropin hormones ("microdose flare protocol"), an oocyte collection procedure and a single embryo transfer.

The patient population will be randomized using computer-generated random table into three arms:

* Luteal Phase Arm: LEI in mid-luteal phase (day 21-26) prior to the treatment cycle.
* Proliferative Phase Arm: LEI in early proliferative phase of current treatment cycle (day 2-3).
* Control Arm: No LEI will be performed. Patients will undergo a routine fresh IVF treatment cycle.

Other than the local endometrial injury, all patients will receive the same treatment and follow up care as per standard practice at our clinic.

All patients in this study will undergo a "microdose flare protocol" fresh IVF cycle. As part of this protocol patients are to take oral contraception pills for a month duration prior to the start of the IVF cycle. Therefore the possibility of an undocumented pregnancy at the time of the LEI in the luteal phase is minimized.

The LEI will be performed using the standard technique using a Pipelle sampling catheter in the outpatient department. After a speculum examination is performed and the cervix is well visualized, the Pipelle will be inserted gently through the cervical canal into the uterine cavity and advanced slowly until resistance is noted. At this point the internal piston is withdrawn to create negative suction and the Pipelle is gently maneuvered up and down alongside the uterine cavity wall. The Pipelle catheter is then withdrawn gently and any obtained specimen (uterine lining) will be sent for histopathological examination.

Both the embryologist who prepares the embryo and the physician who will transfer the embryo will not be directly aware of which study arm the patient was allocated to. However all procedures performed at our clinic, including a LEI, are documented on the patients chart and therefore are accessible.

As per routine practice at our clinic, pregnancy tests will be performed by quantitative serum beta-hCG level 12 days after embryo transfer. A clinical pregnancy will be confirmed by using a transvaginal ultrasound 2 weeks after a positive pregnancy test (serum BHCG).

ELIGIBILITY:
Inclusion Criteria:

* Infertile patients age ≥36 years old.
* Patients who are planned to undergo a second fresh IVF cycle
* Patients who have previously had a fresh IVF-ET and ≥1 frozen - thawed ET in the past and did not achieve a clinical pregnancy [two or more failed embryo transfers].
* Ovarian stimulation with a "microdose flare" protocol
* Patients who are scheduled to undergo a single embryo transfer
* Consent in writing to participate in the study.

Exclusion Criteria:

* Age of <36 years old.
* Known or suspected intrauterine factor on ultrasound imaging (submucosal fibroid, endometrial polyp, intrauterine adhesions or intramural fibroids causing uterine distortion).
* Endometriosis (documented by laparoscopy or known endometriomas by ultrasound)
* Previous hysteroscopy (since the start of their 1st IVF cycle)
* Patients who does not speak English or French.
* Patients who will be transferred more than one embryo.

Ages: 36 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 360 (Estimated)
Dates: Start 2013-08; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Implantation Rate | 4-5 weeks after embryo transfer
  Implantation rate is defined as the number of intrauterine gestational sacs seen on transvaginal ultrasound (clinical pregnancy) divided by the number of embryos transferred [implantation rate = number of gestational sacs noted on the viability ultrasound / number of embryos transferred].

SECONDARY OUTCOMES:
biochemical pregnancy rate | 2 weeks after embryo transfer
  Blood test = BHCG
clinical pregnancy rate | 4-6 weeks after embryo transfer
  A clinical pregnancy is defined as the presence of an intrauterine embryo with fetal heart rate seen on transvaginal ultrasound.
Live birth rate | within 1 year of embryo transfer
  A live birth is defined as having a delivery of a baby >20 weeks gestational age and birth weight >500grams.
Miscarriage Rates | Within 5 months of embryo transfer
  A clinical miscarriage (gestational age <20weeks or birthweight <500g)

CONTACTS AND LOCATIONS:
Overall Officials: Dan Nayot, BSc; MSc; MD, Study Director — McGill University Health Centre/Research Institute of the McGill University Health Centre; Togas Tulandi, MD, MHCM, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Hananel Holzer, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada